CLINICAL TRIAL: NCT00991328
Title: Tailored Patient Management Guided With Absolute Cerebral Oximetry to Prevent Neurocognitive Injury in Elderly Patients Undergoing Cardiac Surgery.
Brief Title: Role of Absolute Cerebral Oximetry to Prevent Neurocognitive Injury in Elderly Patients Undergoing Cardiac Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low enrollment
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GCO # 07-0332
Record Dates: First submitted 2009-10-02; First posted 2009-10-08 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Post-Operative Delirium; Postoperative Cognitive Dysfunction
Keywords: PD; POCD; Post-op Delirium (PD); Post-op Cognitive Dysfunction (POCD)
MeSH Terms: conditions — Emergence Delirium; Postoperative Cognitive Complications

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cerebral Desaturation, i.e; SctO2 < 60 % for 5 minutes (Active Comparator): Once the cerebral desaturation is established, the study personnel will attempt to optimize the level of oxygen within the brain of the study patients.
  Interventions: Procedure: SctO2 < 60 %.
- Patients with SctO2 less than 60 %. (No Intervention): The study patients will not get any intervention in this arm if the Sct02 falls below 60%

INTERVENTIONS:
Procedure: SctO2 < 60 %. — The following intervention protocol will be applied when SctO2 level falls below 60 %. First, the patients head position will be checked for suitable position and the face will be observed for plethora. Then the efforts will be made to maintain PaCO2 between 40-50 mmHg and MAP of 60 - 80 mm Hg. Cardiac index will be maintained between 2.0 - 2.5 L/min/m2. The hematocrit should be more than 20 %. The red blood cells or hemoconcentration will be used for this purpose.
  Arms: Cerebral Desaturation, i.e; SctO2 < 60 % for 5 minutes

SUMMARY:
The purpose of this study is to determine whether brain oxygenation measured by cerebral oximeter has an impact on neurocognitive dysfunction.

DETAILED DESCRIPTION:
Both postoperative delirium (PD) and postoperative cognitive dysfunction (POCD) are well known complications seen in elderly patients after cardiac surgery. The etiologies of PD and POCD are unknown, but cerebral ischemia remains a prime candidate. Attempts to correlate reduced levels of systemic oxygenation (i.e. SpO2) with the development of PD/POCD have been to date disappointing.

We believe that cerebral oximetry, a noninvasive technology that continuously monitors cerebral tissue oxygen saturation (SctO2), will enable us to answer the question of whether or not a correlation exists.

The availability of an absolute cerebral oximeter (FORE-SIGHT), with its ability to establish and manipulate threshold values for SctO2, provides us the opportunity to assess the relationship between cerebral oxygenation and the development of neurocognitive complications.

We propose a randomized, masked trial of 120 patients, adequately powered to assess the following:

* Is there an association between deficits in cerebral oxygenation and the occurrence of PD at some time in the 1st 5 days after the operation?
* Is there an association between deficits in cerebral oxygenation and changes in POCD scores shortly (5 days) after the operation and/or 4-6 weeks later? We hypothesize that individually tailored patient management guided with intraoperative and postoperative absolute cerebral oximetry monitoring using a tailored protocol designed to maintain SctO2 values above a specific threshold will result in improved neurocognitive outcomes in geriatric patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* 65 and older
* Elective cardiac or thoracic aortic surgery
* Capable and willing to consent
* Participants literate in English

Exclusion Criteria:

* Emergency Surgery
* Major Neurological Disease
* Gross Cognitive Dysfunction
* Patients not expected to be able to complete the 1 week and 3 months post-operative visit.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The association of Postoperative Delirium (PD) and Postoperative Cognitive Dysfunction (POCD) with changes in cerebral tissue oxygen saturation (SctO2). | First 5 days after the cardiac surgery.

SECONDARY OUTCOMES:
Postoperative Morbidity and Mortality | 3 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Fischer, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Roach GW, Kanchuger M, Mangano CM, Newman M, Nussmeier N, Wolman R, Aggarwal A, Marschall K, Graham SH, Ley C. Adverse cerebral outcomes after coronary bypass surgery. Multicenter Study of Perioperative Ischemia Research Group and the Ischemia Research and Education Foundation Investigators. N Engl J Med. 1996 Dec 19;335(25):1857-63. doi: 10.1056/NEJM199612193352501. PMID 8948560
- [Background] Newman MF, Kirchner JL, Phillips-Bute B, Gaver V, Grocott H, Jones RH, Mark DB, Reves JG, Blumenthal JA; Neurological Outcome Research Group and the Cardiothoracic Anesthesiology Research Endeavors Investigators. Longitudinal assessment of neurocognitive function after coronary-artery bypass surgery. N Engl J Med. 2001 Feb 8;344(6):395-402. doi: 10.1056/NEJM200102083440601. PMID 11172175
- [Background] Warner CD, Weintraub WS, Craver JM, Jones EL, Gott JP, Guyton RA. Effect of cardiac surgery patient characteristics on patient outcomes from 1981 through 1995. Circulation. 1997 Sep 2;96(5):1575-9. doi: 10.1161/01.cir.96.5.1575. PMID 9315549
- [Background] Inouye SK. Delirium in older persons. N Engl J Med. 2006 Mar 16;354(11):1157-65. doi: 10.1056/NEJMra052321. No abstract available. PMID 16540616
- [Background] Newman MF, Grocott HP, Mathew JP, White WD, Landolfo K, Reves JG, Laskowitz DT, Mark DB, Blumenthal JA; Neurologic Outcome Research Group and the Cardiothoracic Anesthesia Research Endeavors (CARE) Investigators of the Duke Heart Center. Report of the substudy assessing the impact of neurocognitive function on quality of life 5 years after cardiac surgery. Stroke. 2001 Dec 1;32(12):2874-81. doi: 10.1161/hs1201.099803. PMID 11739990
- [Background] Ergin MA, Galla JD, Lansman sL, Quintana C, Bodian C, Griepp RB. Hypothermic circulatory arrest in operations on the thoracic aorta. Determinants of operative mortality and neurologic outcome. J Thorac Cardiovasc Surg. 1994 Mar;107(3):788-97; discussion 797-9. PMID 8127108
- [Background] Plestis KA, Gold JP. Importance of blood pressure regulation in maintaining adequate tissue perfusion during cardiopulmonary bypass. Semin Thorac Cardiovasc Surg. 2001 Apr;13(2):170-5. doi: 10.1053/stcs.2001.24071. PMID 11494208
- [Background] Hagl C, Khaladj N, Karck M, Kallenbach K, Leyh R, Winterhalter M, Haverich A. Hypothermic circulatory arrest during ascending and aortic arch surgery: the theoretical impact of different cerebral perfusion techniques and other methods of cerebral protection. Eur J Cardiothorac Surg. 2003 Sep;24(3):371-8. doi: 10.1016/s1010-7940(03)00337-3. PMID 12965307
- [Background] Rasmussen LS, O'Brien JT, Silverstein JH, Johnson TW, Siersma VD, Canet J, Jolles J, Hanning CD, Kuipers HM, Abildstrom H, Papaioannou A, Raeder J, Yli-Hankala A, Sneyd JR, Munoz L, Moller JT; ISPOCD2 Investigators. Is peri-operative cortisol secretion related to post-operative cognitive dysfunction? Acta Anaesthesiol Scand. 2005 Oct;49(9):1225-31. doi: 10.1111/j.1399-6576.2005.00791.x. PMID 16146456
- [Background] Goldman S, Sutter F, Ferdinand F, Trace C. Optimizing intraoperative cerebral oxygen delivery using noninvasive cerebral oximetry decreases the incidence of stroke for cardiac surgical patients. Heart Surg Forum. 2004;7(5):E376-81. doi: 10.1532/HSF98.20041062. PMID 15799908
- [Background] Murkin JM, Adams SJ, Novick RJ, Quantz M, Bainbridge D, Iglesias I, Cleland A, Schaefer B, Irwin B, Fox S. Monitoring brain oxygen saturation during coronary bypass surgery: a randomized, prospective study. Anesth Analg. 2007 Jan;104(1):51-8. doi: 10.1213/01.ane.0000246814.29362.f4. PMID 17179242
- [Background] Moller JT, Cluitmans P, Rasmussen LS, Houx P, Rasmussen H, Canet J, Rabbitt P, Jolles J, Larsen K, Hanning CD, Langeron O, Johnson T, Lauven PM, Kristensen PA, Biedler A, van Beem H, Fraidakis O, Silverstein JH, Beneken JE, Gravenstein JS. Long-term postoperative cognitive dysfunction in the elderly ISPOCD1 study. ISPOCD investigators. International Study of Post-Operative Cognitive Dysfunction. Lancet. 1998 Mar 21;351(9106):857-61. doi: 10.1016/s0140-6736(97)07382-0. PMID 9525362
- [Background] Murkin JM. Hemodynamic changes during cardiac manipulation in off-CPB surgery: relevance in brain perfusion. Heart Surg Forum. 2002;5(3):221-4. PMID 12538133
- [Background] Ferrari M, Mottola L, Quaresima V. Principles, techniques, and limitations of near infrared spectroscopy. Can J Appl Physiol. 2004 Aug;29(4):463-87. doi: 10.1139/h04-031. PMID 15328595
- [Background] Madsen PL, Secher NH. Near-infrared oximetry of the brain. Prog Neurobiol. 1999 Aug;58(6):541-60. doi: 10.1016/s0301-0082(98)00093-8. PMID 10408656
- [Background] Yao FS, Tseng CC, Ho CY, Levin SK, Illner P. Cerebral oxygen desaturation is associated with early postoperative neuropsychological dysfunction in patients undergoing cardiac surgery. J Cardiothorac Vasc Anesth. 2004 Oct;18(5):552-8. doi: 10.1053/j.jvca.2004.07.007. PMID 15578464
- [Background] Moraca R, Lin E, Holmes JH 4th, Fordyce D, Campbell W, Ditkoff M, Hill M, Guyton S, Paull D, Hall RA. Impaired baseline regional cerebral perfusion in patients referred for coronary artery bypass. J Thorac Cardiovasc Surg. 2006 Mar;131(3):540-6. doi: 10.1016/j.jtcvs.2005.10.046. Epub 2006 Jan 31. PMID 16515903
- [Background] Nakamura Y, Kawachi K, Imagawa H, Hamada Y, Takano S, Tsunooka N, Sugishita H, Sakoh M. The prevalence and severity of cerebrovascular disease in patients undergoing cardiovascular surgery. Ann Thorac Cardiovasc Surg. 2004 Apr;10(2):81-4. PMID 15209548
- [Background] Reents W, Muellges W, Franke D, Babin-Ebell J, Elert O. Cerebral oxygen saturation assessed by near-infrared spectroscopy during coronary artery bypass grafting and early postoperative cognitive function. Ann Thorac Surg. 2002 Jul;74(1):109-14. doi: 10.1016/s0003-4975(02)03618-4. PMID 12118739
- [Background] Oki A, Ohtake H, Okada Y, Kawada T, Takaba T. Simultaneous monitoring of somatosensory evoked potentials and regional cerebral oxygen saturation combined with serial measurement of plasma levels of cerebral specific proteins for the early diagnosis of postoperative brain damage in cardiovascular surgery. J Artif Organs. 2004;7(1):13-8. doi: 10.1007/s10047-003-0242-8. PMID 15083339
- [Background] Ito H, Kanno I, Fukuda H. Human cerebral circulation: positron emission tomography studies. Ann Nucl Med. 2005 Apr;19(2):65-74. doi: 10.1007/BF03027383. PMID 15909484
- [Background] Macmillan CS, Andrews PJ. Cerebrovenous oxygen saturation monitoring: practical considerations and clinical relevance. Intensive Care Med. 2000 Aug;26(8):1028-36. doi: 10.1007/s001340051315. PMID 11030158
- [Background] Grocott HP, Mackensen GB, Grigore AM, Mathew J, Reves JG, Phillips-Bute B, Smith PK, Newman MF; Neurologic Outcome Research Group (NORG); Cardiothoracic Anesthesiology Research Endeavors (CARE) Investigators' of the Duke Heart Center. Postoperative hyperthermia is associated with cognitive dysfunction after coronary artery bypass graft surgery. Stroke. 2002 Feb;33(2):537-41. doi: 10.1161/hs0202.102600. PMID 11823666
- [Background] Souter MJ, Andrews PJ, Alston RP. Jugular venous desaturation following cardiac surgery. Br J Anaesth. 1998 Aug;81(2):239-41. doi: 10.1093/bja/81.2.239. PMID 9813529
- [Background] Raymond TL, Lofland HB, Clarkson TB. Cholesterol metabolism in squirrel monkeys: analysis of long-term kinetic studies in plasma and body tissues. Exp Mol Pathol. 1976 Dec;25(3):344-54. doi: 10.1016/0014-4800(76)90044-7. No abstract available. PMID 826406
- [Background] Marcantonio ER, Juarez G, Goldman L, Mangione CM, Ludwig LE, Lind L, Katz N, Cook EF, Orav EJ, Lee TH. The relationship of postoperative delirium with psychoactive medications. JAMA. 1994 Nov 16;272(19):1518-22. PMID 7966844